CLINICAL TRIAL: NCT01542242
Title: Liraglutide Use in Prader-Willi Syndrome
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Subject withdrew
Sponsor: Vancouver General Hospital (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, David E. Harris, MD, MD, Clinical Endocrinology Fellow, University of British Columbia, Vancouver General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PWS.VGH.UBC
Record Dates: First submitted 2012-02-21; First posted 2012-03-02 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes Mellitus Type 2; Prader Willi Syndrome
Keywords: Diabetes Mellitus Type 2; Prader Willi Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prader-Willi Syndrome | interventions — Liraglutide

ARMS (1):
- Liraglutide (Experimental): Treatment of Diabetes Mellitus Type 2 with Liraglutide in the setting of Prader Willi Syndrome
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Liraglutide 0.6 mg SQ daily for one week, increase to a maximum dose of 1.8 mg SQ daily by 6 weeks, and subsequent continuation for the remainder of a year.
  Other Names: Victoza

SUMMARY:
Liraglutide is a glucagon like peptide -1 (GLP-1) agonist, which is approved for use in patients with type 2 diabetes. Studies of liraglutide have shown an appetite suppressive effect and has been associated with weight loss in patients with type 2 diabetes. Liraglutide use in the treatment of PWS is limited to one case report by Cyganek et el (See attached Citation). In this case report, the subject showed improvements in hemoglobin A1c and body weight over 14 weeks.

The investigators plan to examine the use of liraglutide in a single subject with Prader Willi Syndrome and type 2 diabetes for one year. The investigators will examine clinical parameters, clinical assessment of hunger, and biochemical markers of diabetes and lipid control.

ELIGIBILITY:
Inclusion Criteria:

* Prader Willi Syndrome, Diabetes Type 2

Exclusion Criteria:

* Previous or family history of Medullary Carcinoma of the Thyroid or multiple endocrine neoplasia syndrome.
* Subjects with acute or chronic Pancreatitis

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C | Change from baseline in A1C at 12 months

SECONDARY OUTCOMES:
Fasting Blood Glucose (mmol/L) | Change from baseline in fasting blood glucose at 12 months
Fasting Blood Insulin level | Change from baseline in fasting blood insulin at 12 months
Body Weight (kg) | Change from baseline in body weight at 12 months
Fasting Lipid Profile | Change from baseline in fasting lipid profile at 12 months
Hip Circumference (cm) | Change from baseline in hip circumference at 12 months
Total Body Adipose Tissue Distribution (whole body Computed Tomography) | Change from baseline in total body adipose tissue distribution at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jason Kong, MD, FRCPC, Principal Investigator — Vancouver General Hospital, University of British Columbia
Locations (1):
- Vancouver General Hospital - Diamond Center, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Cyganek K, Koblik T, Kozek E, Wojcik M, Starzyk J, Malecki MT. Liraglutide therapy in Prader-Willi syndrome. Diabet Med. 2011 Jun;28(6):755-6. doi: 10.1111/j.1464-5491.2011.03280.x. No abstract available. PMID 21388446
- [Background] Sze L, Purtell L, Jenkins A, Loughnan G, Smith E, Herzog H, Sainsbury A, Steinbeck K, Campbell LV, Viardot A. Effects of a single dose of exenatide on appetite, gut hormones, and glucose homeostasis in adults with Prader-Willi syndrome. J Clin Endocrinol Metab. 2011 Aug;96(8):E1314-9. doi: 10.1210/jc.2011-0038. Epub 2011 Jun 1. PMID 21632815